CLINICAL TRIAL: NCT00283725
Title: Review of Management Strategies in Dementia
Brief Title: Use of Different Treatment Care Methods in Patients With Dementia Associated With Alzheimer's Disease
Acronym: REMIND
Status: Completed | Type: Observational
Sponsor: Ortho-McNeil Neurologics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR004636; GALALZ4004 (Other: Ortho-McNeil Neurologics, Inc.); GAL-OUT-065 (Other: Ortho-McNeil Neurologics, Inc.); NCT01712932 (obsolete NCT alias)
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Dementia; Alzheimer's Disease
Keywords: Dementia; Alzheimer's Disease; Acetylcholinesterase inhibitor; Galantamine; Nursing Home Admission
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Galantamine
  Interventions: Other: No intervention
- No Alzheimer's disease (AD) treatment
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Patients will be prescribed either galantamine or no AD treatment (ie, neither an acetylcholinesterase inhibitor [AChEI] nor memantine).

SUMMARY:
The purpose of this observational study is to examine patterns of treatment care for patients with Alzheimer's disease (AD) in a real-world arena and to examine the association with different outcomes for patients and informal caregivers.

DETAILED DESCRIPTION:
This is a 2-year, multicenter, prospective (look forward using periodic observations collected predominantly following patient enrollment), longitudinal (it is a co relational research study that involves repeated observations of the same variables over long periods of time), and observational study. The objective of this study is to examine the patients with mild and moderate AD who are currently being treated with different treatment care methods in real-world settings. Doctors will not be provided medication or asked to treat their patients with any particular treatment. The effect of the different management strategies on cognition, activities of daily living, and behavior of the patients will be evaluated, and data on the informal caregiver burden will be assessed. Data on the utilization of health and social care services by the patient and the primary informal caregiver, including admission of the patient to an assisted living facility or nursing home will be assessed. The doctor's assessment of clinical global impression and adverse events will also be documented. Data will be collected from the doctors at baseline and at 6, 12, and 24 months, and from the caregivers at baseline and 6, 12, 18, and 24 months. The medication dosage and administration is based upon the doctors' prescription, individualized for the patient and not dictated by the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Have a physician-based diagnosis of mild to moderate Alzheimer's disease (Mini-Mental State Examination [MMSE] score between 10-24)
* Must be living at home or in a facility for the elderly (eg, assisted living), who live with or have frequent visits from a friend or relative (caregiver) or with a behavioral symptom (eg, as agitation or wandering)
* Have no plan to change the current treatment plan for at least 90 days

Exclusion Criteria:

* Have been using an acetylcholinesterase inhibitor or memantine currently but have used one in the past 30 days
* Must be residing in or planning to move to a nursing home within the next 90 days or patients participating in another clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with demetia with mild to moderate Alzheimer's disease.
Sampling Method: Non-Probability Sample
Enrollment: 573 (Actual)
Dates: Start 2003-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Mini Mental State Examination (MMSE) scale score at Month 24 | Baseline, Month 24
  MMSE is a brief 30-point questionnaire test that is used for the assessment of dementia patients' cognitive impairment. Evaluation of points are as: 24-30 = No cognitive impairment, 18-23 = Mild cognitive impairment, 0-17 = Severe cognitive impairment. Lower scores indicate worsening.

SECONDARY OUTCOMES:
Change from baseline in clinical global impression (CGI) scale score at Month 24 | Baseline, Month 24
  The CGI rating scale is a 7-point global assessment that measures the clinician's impression of the severity of illness exhibited by a patient. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill patients". Higher scores indicate worsening.
Change from baseline in Neuropsychiatric Inventory Questionnaire (NPI-Q) at Month 24 | Baseline, Month 24
  The NPI is a validated clinical instrument for evaluating psychopathology in dementia to quantify and qualitate changes in psychiatric symptoms. It has 13-point scale and each is rated as follows: 1= mild (noticeable, but not a significant change), 2= moderate (significant, but not a dramatic change), and 3= Severe (very marked and prominent: a dramatic change). Higher scores indicate worsening.
Change from baseline in Zarit caregiver burden scale score at Month 24 | Baseline, Month 24
  Zarit caregiver burden scale is used to measure caregiver burden as it relates to time, developmental comparison with peers, physical health, social relationships, and emotional health. It has 22 item and each question is scored on a 5-point Likert scale ranging from 0 = never present to 4 = nearly always present. The sum of the total scores of the 22-items is calculated in the range from 0 (low burden) to 88 (high burden). Higher scores indicate worsening.
Change from baseline in Kaplan-Meier estimate at Month 24 | Baseline, Month 24
  By using Kaplan-Meier Estimator, the effect of an intervention is assessed by measuring the number of patients survived or saved after that intervention is given over a period of time. At any time point, the survival will be measured by the following formula: Number of patients living at the start minus Number of patients died divided by Number of patients living at the start.
Number of patients with adverse events | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Neurologics, Inc. Clinical Trial, Study Director — Ortho-McNeil Neurologics, Inc.

REFERENCES:
- See also: Review of Management Strategies in dementia -REMIND — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=918&filename=CR004636_CSR.pdf